CLINICAL TRIAL: NCT00618826
Title: A Phase II Trial of Biweekly Gemcitabine, Paclitaxel, and Avastin as Frontline Therapy for Metastatic Breast Cancer
Brief Title: A Study of Biweekly Gemcitabine, Paclitaxel, and Avastin in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Sayeh Lavasani, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-050; 2007-050 (Other: Barbara Ann Karmanos Cancer Institute); B9E-US-I158 (Other: Eli Lilly); AVF3734s (Other: Genentech)
Record Dates: First submitted 2008-02-07; First posted 2008-02-20 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Gemcitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Period (Experimental): Treatment will be administered once every 2 weeks. One cycle of therapy will consist of 14 days. Paclitaxel is administered first after appropriate premedications. Gemcitabine is administered second and Avastin is administered after chemotherapy, all given on day 1 of each cycle.
  Interventions: Drug: Paclitaxel; Drug: Gemcitabine; Drug: Avastin

INTERVENTIONS:
Drug: Paclitaxel — Patients will be premedicated with dexamethasone and diphenhydramine hydrochloride. Patients will received 150mg of paclitaxel via IV over 120 mins.
Drug: Gemcitabine — Patients will receive 1500mg of Gemcitabine via IV over 30-60 minutes. Gemcitabine will be given after Paclitaxel.
Drug: Avastin — 10mg/kg will be given via IV over 90 mins (1st dose). Patients must remain under supervision for 1 hr after completion of the initial dose of Avastin. If no side effects occur, shortened, 60-min 2nd infusion, the post-infusion observation period for the subsequent infusions may be shortened to 20 minutes, and eliminated entirely with the fourth and subsequent infusions.

SUMMARY:
The purpose of this study is to look at a new chemotherapy schedule in metastatic breast cancer.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether a new chemotherapy schedule using biweekly combination of paclitaxel (Taxol®), gemcitabine (Gemzar®) and Avastin would help to lessen in-between-cycle growth of resistant cells and to evaluate the toxicity of this therapy.

Taxol is approved by the Food and Drug Administration (FDA) for use in metastatic breast and metastatic ovarian cancer but its use in this study is investigational. Gemzar is FDA approved for the use in breast, lung and pancreatic cancer but its use in this study is investigational.

The Avastin being given in this study is commercially available, however, it has not been approved by FDA for use in metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older with histologically confirmed breast cancer and clinical evidence of metastatic disease.
* Patients must have measurable or non-measurable disease. X-rays, scans or physical examinations used to assess measurable disease must be performed within 28 days prior to registration. X-rays, scans or physical examinations to assess non-measurable disease must be completed within 42 days prior to registration. Patients with effusions or ascites as the only sites of disease are ineligible.
* Patients must meet the following requirements regarding prior and concurrent chemotherapy:Patients must not have received prior chemotherapy regimens for metastatic breast cancer. Patients may have received adjuvant/neoadjuvant chemotherapy, for a total of 3 prior regimens.
* Prior therapy with paclitaxel or docetaxel is allowed in the adjuvant or neoadjuvant setting, if given > 6 months prior to registration.
* Patients must have >14 days delay between the conclusion of any radiation and the start of gemcitabine, provided the acute effects of radiation treatment have resolved.
* Patients may have received any number of exogenous hormonal therapies and/or trastuzumab in the adjuvant, neoadjuvant or metastatic setting. Last dose of prior hormonal therapy at least 14 days prior to registration.
* Patients may receive concomitant bisphosphonate therapy for bone metastasis.
* Patients must have recovered from any prior surgery. Two weeks must have elapsed from the time of any minor surgery and 4 weeks of any major surgery.
* Patients must have adequate bone marrow reserve as evidenced by the following: ANC > 1500/mcL, platelets > 100, 000/mcL, and hemoglobin > 9.0 gm/dL. These results must be obtained within 28 days prior to registration.
* Patients must have serum creatinine < 1.5 mg/dL, obtained within 28 days prior to registration.
* Urine Protein: creatinine ratio ≥ 1.0 at screening.
* Patients must have adequate liver function.
* Patients must have a Zubrod performance status of 0-1.

Exclusion Criteria:

* Patients must not have tumors that carry HER-2 gene amplifications as determined by (i) fluorescence in situ hybridization (FISH) or (ii) overexpression of HER-2 protein 3+ level assessed by immunohistochemistry; or may have tumors that carry HER=2 gene amplification and have had disease progression while on trastuzumab. Patients who have previously been treated with trastuzumab must be off treatment at least 28 days prior to registration.
* Patients must not have CNS metastasis, leptomeningeal disease or lymphatic pulmonary metastases.
* Patients must not have had prior therapy with gemcitabine or bevacizumab.
* Patient must not have major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to start of treatment, anticipation of need for major surgical procedure during the course of the study.
* Patients must not have received radiation to > 50% of the marrow-bearing bone.
* Patients must not have a history of significant symptomatic cardiac disease or left ventricular ejection fraction (LVEF) < 50% of the institutional lower limit of normal (ILLN). An isotope cardiac scan (MUGA) and ECG must be obtained within 28 days.
* Patients with uncontrolled hypertension are NOT eligible (BP>150/100).
* Patients must not have pr-existing clinically significant (Grade 2 or greater per CTCAE Version 3.0 motor or sensory neuropathy except for abnormalities due to cancer.
* Patients known to be HIV positive.
* Patients must not be nursing or pregnant. Men and women of reproductive potential must agree to use an effective contraceptive method.
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or Stage II cancer from which the patient has been disease free for 5 years.
* Patients must not have had a Stroke or Myocardial Infarction in the past 6 months. Patients with unstable agina, significant peripheral vascular disease, history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within the last 6 months should be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sayed Lavasani, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel + Gemcitabine + Avastin: Treatment administered once every 2 weeks, 1 cycle will consist of 14 days.
  Paclitaxel (administered first) - Patients will be pre-medicated with dexamethasone and diphenhydramine hydrochloride. Patients will received 150mg of paclitaxel via IV over 120 mins.
  Gemcitabine (given after Paclitaxel) - Patients will receive 1500mg of Gemcitabine via IV over 30-60 minutes. Gemcitabine will be given after Paclitaxel.
  Avastin - 10mg/kg will be given via IV over 90 mins (1st dose). Patients must remain under supervision for 1 hr after completion of the initial dose of Avastin. If no side effects occur, shortened, 60-min 2nd infusion, the post-infusion observation period for the subsequent infusions may be shortened to 20 minutes, and eliminated entirely with the fourth and subsequent infusions.
Period: Overall Study
Arm/Group | Paclitaxel + Gemcitabine + Avastin
Started | 14
Completed | 13
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Period
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 53.5 [34 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Time from study entry to disease progression or death
Time Frame: maximum 50 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Treatment: Paclitaxel / Gemcitabine
Arm/Group | Treatment
Number analyzed (Participants) | 13
months | 43 [7 to 45]

2. Secondary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: maximum 50 months
Population: patients with measurable disease
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Arm 1: all participants
Arm/Group | Arm 1
Number analyzed (Participants) | 13
proportion of participants | 0.46 [0.19 to 0.75]

3. Other Pre Specified Outcome: Overall Survival (OS) at 3 Years
Description: proportion of participants surviving 3 years
Time Frame: 3 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Toxicity
Description: toxicities recorded using CTCAE definitions
Time Frame: Duration of study
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Treatment Period
Serious Adverse Events (participants affected / at risk) | 10/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period (N=14)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2)
Rigors/chills (General disorders) | 1 (1)
Dermatology/Skin-Other (Specify,_) (Skin and subcutaneous tissue disorders) | 1 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils-Skin (cellulitis) (Infections and infestations) | 1 (1)
Infection with unknown ANC - Bronchus (Infections and infestations) | 1 (1)
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1 (3)
Infection with unknown ANC - Upper airway NOS (Infections and infestations) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 1 (1)
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 1 (1)
Glucose, serum-high (hyperglycemia) (Investigations) | 3 (3)
Potassium, serum-high (hyperkalemia) (Investigations) | 1 (2)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (2)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Pain-Extremity-limb (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain-Joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain-Muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain-Pain NOS (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain-Other (Specify,_) (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period (N=14)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 4 (5)
Blood/Bone Marrow - Other (Specify,_) (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 11 (16)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 3 (6)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (2)
Platelets (Blood and lymphatic system disorders) | 10 (13)
Supraventricular and nodal arrhythmia-Sinus tachycardia (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia-Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 5 (5)
Thrombotic microangiopathy (e.g., thrombocytopenic purpura [TTP] or hemolytic uremic syndrome [HUS]) (Blood and lymphatic system disorders) | 1 (1)
Constitutional Symptoms-Other(Specify,_) (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 12 (26)
Fever (in the absense of neutropenia is defined as ANC <1.0 x10e9/L) (General disorders) | 4 (5)
Edema: limb-1 (General disorders) | 3 (3)
Rigors/chills (General disorders) | 4 (4)
Sweating (diaphoresis) (General disorders) | 2 (3)
Weight loss (Investigations) | 5 (5)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (2)
Dermatology/Skin-Other (Specify,_) (Skin and subcutaneous tissue disorders) | 3 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 6 (6)
Nail changes (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash:erythema multiforme (e.g., Steven-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (4)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes/flushes (Endocrine disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 5 (7)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal- Other (Specify,_) (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (clinical exam)-Oral cavity (Gastrointestinal disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 10 (15)
Vomiting (Gastrointestinal disorders) | 8 (12)
Hemorrhage,pulmonary/upper respiratory-Nose (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Hemorrhage/Bleeding - Other (Specify,_) (Gastrointestinal disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hemorrhage, GI-Varices (rectal) (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils-Bronchus (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils-Oral cavity-gums (gingivitis) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 1 (1)
Infection with unknown ANC-Bronchus (Infections and infestations) | 1 (1)
Infection with unknown ANC-Nose (Infections and infestations) | 1 (1)
Infection with unknown ANC-Paranasal (Infections and infestations) | 1 (1)
Infection with unknown ANC-Pharynx (Infections and infestations) | 2 (2)
Infection with unknown ANC-Skin (cellulitis) (Infections and infestations) | 2 (3)
Infection with unknown ANC-Upper airway NOS (Infections and infestations) | 1 (1)
Infection with unknown ANC-Urinary tract NOS (Infections and infestations) | 1 (1)
Infection with unknown ANC-Wound (Infections and infestations) | 1 (1)
Edema: head and neck (General disorders) | 1 (1)
Edema:limb (General disorders) | 3 (3)
Lymphedema-related fibrosis (Vascular disorders) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Investigations) | 1 (1)
Alkaline phosphatase (Investigations) | 5 (6)
ALT,SGPT (serum glutamic pyruvic transaminase) (Investigations) | 5 (7)
AST,SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 6 (6)
Bilirubin(hyperbilirubinemia) (Investigations) | 1 (1)
Calcium, serum-high (hypercalcemia) (Investigations) | 1 (1)
Calcium, serum-low (hypocalcemia) (Investigations) | 1 (1)
Creatinine (Investigations) | 2 (3)
Glucose, serum-high (hyperglycemia) (Investigations) | 12 (23)
Glucose, serum-low (hypoglycemia) (Investigations) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Investigations) | 1 (1)
Metabolic/Laboratory - Other (Specify,_) (Investigations) | 2 (2)
Potassium, serum-high (hyperkalemia) (Investigations) | 1 (1)
Potassium, serum-low (hypokalemia) (Investigations) | 1 (1)
Proteinuria (Investigations) | 7 (16)
Sodium, serum-low (hyponatremia) (Investigations) | 2 (2)
Uric acid, serum-high (hyperuricemia) (Investigations) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Mood alteration-Anxiety (Nervous system disorders) | 3 (3)
Mood alteration-Depression (Nervous system disorders) | 2 (2)
Neurology- Other(Specify,_) (Nervous system disorders) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 10 (19)
Dry eye syndrome (Eye disorders) | 1 (1)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 4 (4)
Vision-flashing lights/floaters (Eye disorders) | 1 (1)
Pain-Back (Musculoskeletal and connective tissue disorders) | 4 (7)
Pain-Bone (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain-Chest wall (Musculoskeletal and connective tissue disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pain-External ear (Ear and labyrinth disorders) | 1 (1)
Pain-Extremity-limb (Musculoskeletal and connective tissue disorders) | 5 (6)
Pain-Face (General disorders) | 1 (1)
Pain-Head/headache (General disorders) | 3 (3)
Pain-Joint (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain (General disorders) | 1 (1)
Pain-Muscle (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain-Pain NOS (General disorders) | 6 (7)
Pain-Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pain-Other (Specify,_) (General disorders) | 1 (2)
Bronchospasm,wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory-Other (Specify,_) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Voice changes/dysarthria (e.g. hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 1 (1)
Renal/Genitourinary-Other(Specify,_) (Renal and urinary disorders) | 2 (3)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Vaginal mucositis (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No